CLINICAL TRIAL: NCT04121624
Title: A New Mobile Phone Application for Blood Pressure Monitoring: A Comparison With the Oscillometric Brachial Cuff in Patients Treated in The Emergency Department
Brief Title: Evaluation of a Novel Mobile Phone Application ( OptiBP) for Blood Pressure Monitoring
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, MD PhD, Principal Investigator, Erasme University Hospital
Other Study IDs: P2019/375
Record Dates: First submitted 2019-10-03; First posted 2019-10-10 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Technology
MeSH Terms: interventions — Blood Pressure Monitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: novel mobile phone application for blood pressure monitoring. — Comparative blood pressure measurement with the smartphone application and the non-invasive reference method (upper arm cuff).

SUMMARY:
Evaluation of a novel smartphone application designed to estimate blood pressure (systolic-diastolic and mean arterial pressure) and heart rate based on collected optical signals on patient's finger treated in the emergency department against the reference method (the oscillometric brachial cuff )

DETAILED DESCRIPTION:
The purpose of the study is to compare the blood pressure values measured by a novel smartphone application ( camera of the smartphone will be obstructed by the patient's right index) and the values measured by reference method used (the oscillometric brachial cuff).

All patients admitted to the emergency department at Erasme Hospital Brussels, Belgium during 5 consecutive weeks will be recruited and their pressure will be measured with both mesurement methods. (novel smartphone application versus upper arm cuff oscillometry).

The OptiBP Application is a mobile application installed on a smartphone which is a non-invasive data-logger intended to acquire physiological data from patients. By applying the patient's finger on a smartphone's camera, a movie is generated and transformed into values of diastolic, mean and systolic blood pressure (+ heart rate), as well as patient's heart rate.

After having compared that the blood pressure in both arms are similar ( maximum of 10 mmHg of blood pressure difference between both arms), three measures will be taken (spaced by one minute) with both methods after a period of 3 minutes of rest (supine position).

The patient's blood pressure will be measured in parallel with the mobile application and with the reference equipment (the oscillometric brachial cuff).

Then, the values obtained by the two methods will be compared to confirm the reliability of the data obtained with the novel mobile application.

The goal is therefore to compare blood pressure values as obtained by the analysis of the data recorded by the OptiBP Mobile Application, against simultaneous measurements provided by the oscillometric brachial cuff

ELIGIBILITY:
Inclusion Criteria:

* Patients (Men or women) older than 18 years old admitted to the emergency department and in relatively good conditions to be able to participate in the study.
* Informed Consent as documented by signature

Exclusion Criteria:

* Minor patients
* Patients unable to participate due to the illness.
* Patients that cannot sign informed consent
* Patients extremely painful at the arrival (not possible for him to stay in a supine position).
* Blood pressure difference between the two arms >10mmHg
* Unstable patients requiring an urgent management

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the Emergency department at Erasme hospital during one month (October 7 th until November 7 th 2019)
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Confirmation of Blood pressure values measured simultanuously with the novel smartphone application | during a 6 minutes period of time in the emergency department.
  Comparision of values to non-invasive reference method (the oscillometric brachial cuff )

SECONDARY OUTCOMES:
Usability assessment | during a 6 minutes period of time in the emergency department.
  Identification of possible use error in the manipulation of the device and in the performance of the measure (finger position, contact pressure, etc).

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre J Joosten, MD PhD, Principal Investigator — ERASME
Locations (1):
- Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Desebbe O, Tighenifi A, Jacobs A, Toubal L, Zekhini Y, Chirnoaga D, Collange V, Alexander B, Knebel JF, Schoettker P, Joosten A. Evaluation of a novel mobile phone application for blood pressure monitoring: a proof of concept study. J Clin Monit Comput. 2022 Aug;36(4):1147-1153. doi: 10.1007/s10877-021-00749-2. Epub 2021 Aug 18. PMID 34409513